CLINICAL TRIAL: NCT01487902
Title: Randomized Phase II Screening Trial of Docetaxel Plus Prednisolone With or Without Androgen Deprivation Treatment in Castrate-Resistant Prostatic Cancer
Brief Title: The Role of Androgen Deprivation Treatment (ADT) in Docetaxe-Prednisolone Chemotherapy for Castrate-Resistant Prostatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOSG-AMC-0803
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Chemotherapy-naive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADT arm (Experimental): Concomitant androgen deprivation treatment
  Interventions: Drug: ADT
- No ADT arm (Active Comparator): No concomitant androgen deprivation treatment arm
  Interventions: Drug: No ADT

INTERVENTIONS:
Drug: ADT — Luprolide 11.25 mg long-acting depo (Lucrin Depot PDS inj®) every 12 weeks SC wit Docetaxel-prednisolone (TAX327 regimen)
  Arms: ADT arm
Drug: No ADT — Docetaxel-prednisolone (TAX327 regimen) alone
  Arms: No ADT arm

SUMMARY:
The purpose of this study is to assess the androgen deprivation therapy when patients with castration-resistant prostate cancer are treated with docetaxel-based chemotherapy.

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) has been the mainstay in the treatment of metastatic prostate carcinoma. Despite initial favorable responses, predictable and irreversible resistance to ADT will occur in the vast majority of patients, which is defined as Castrate-Resistant prostate cancer (CRPC).

Recently, TAX327 study revealed docetaxel plus prednisolone could not only improve the QOL and PSA response but also prolong the survival in CRPC. It has been reasoned that discontinuation of ADT in nonorchiectomized patients may have detrimental effect on patients with CRPC as discontinuation of ADT can result in renewed release of testosterone and possible stimulation of remaining androgen-sensitive elements. When exogenous testosterone therapy is administered to patients with symptomatic CRPC, adverse responses can be induced. However, the lowest concentration of endogenous androgens that is capable of stimulating tumor growth is unknown. Data from animal models of androgen-dependent tumors showed that androgen-independent status is usually followed by androgen-insensitivity, which support the no need for ADT in CRPC. Contradictory, Dunning rat prostate cancer model cell lines, which are androgen-insensitive in vitro and grow slowly in the castrate rat, can grow more rapidly in a host with intact testis. In the retrospective observational study of CRPC treated with anthracycline, platinum, or ketoconazole, Taylor, et al. showed a modest, but statistically significant, survival advantage when ADT is continued. But, Hussain et al. and our team reported that there was no obvious advantage of continued ADT in response to cytotoxic chemotherapy or survival for in patients with CRPC. In addition, prospective trial conducted by Shamash, et al. showed that hormonal sensitivity can be reintroduced by stopping ADT during chemotherapy for CRPC. Among 43 patients who restarted androgen blockade after the completion of chemotherapy without ADT, 37% of patients had PSA response which was associated with survival advantage. Despite the limited and retrospective information available on the impact of continued ADT on disease outcome in CRPC when treated with cytotoxic chemotherapy, especially docetaxel containing regimen, ADT is frequently advocated to be used continuously. Considering little information on the benefit of continued ADT, and cost and side effects of ADT, prospective comparative studies are eagerly needed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Clinical or radiologic evidence of metastatic disease
* Documented disease progression during hormone therapy (ADT with or without antiandrogen)
* Cessation of ADT at least 4 weeks in non-orchiectomized patients
* Adequate duration (at least 4 weeks for flutamide and 6 weeks for bicalutamide) of anti-androgen withdrawal (only for patients who showed a response or decline in PSA for more than 3 months)
* KPS ≥ 60
* No prior cyto-toxic chemotherapy (except estramustine) or radioisotopes
* No prior radiotherapy 25% or more of the bone marrow
* No peripheral neuropathy grade 2 or worse
* Adequate organ and bone marrow function

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Presence or history of CNS metastasis
* Other serious illness or medical conditions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Time to PSA progression | 1 year

SECONDARY OUTCOMES:
Composite progression-free survival (PFS) | 1 year
  PFS based on PSA, RECIST, bone scan, and performance status
Overall survival | 2 year
PSA decline | 12 weeks
PSA response to ADT retrial | 12 weeks
  ADT will be rechallenged to patients assigned to no ADT arm when their disease progress despite of docetaxel-prednisolone chemotherapy.
  The PSA response to ADT rechallenge, such as PSA response based on PCWG v1.0, will be assessed and the number of patients with PSA response and the amount of PSA decline will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Retrospective study on the role of ADT — http://www.ncbi.nlm.nih.gov/pubmed/20686407